CLINICAL TRIAL: NCT00732394
Title: This is a Study is for the Purpose of Quantifying Function of the Back and Lower Extremities, and to Assess the Inter-Regional Biomechanical Relationships of the Neck, Upper Extremities, Back, and Lower Extremities in Patients Suffering From Chronic Low Back Pain.
Brief Title: A Comparative Study: Non-Surgical Spinal Decompression and Spinal Manipulative Therapy- Utilizing a Quantifiable Musculoskeletal Functional Assessment Risk Analysis Tool (MSDR®) in Patients With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MedAppraise, Inc. (Industry)
Responsible Party: Damon J. Stafford, D.C., Back2Life of Florida, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: TCT06-002
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: MSDR — The MSDR® questionnaire establishes an individual's musculoskeletal functional status using information gathered from 1) a questionnaire the patient fills out regarding medical history, chronic medical conditions, and health risk factors; 2) anatomic pain survey completed by the patient; and 3) evaluation by a trained researcher of various patient biometric parameters related to range of motion. Stratifying an individual into a risk category with this evidence-based assessment tool then permits an assessment of which patients respond long term to therapy.
  MSDR® demonstrates the ability to benchmark specific musculoskeletal findings (both clinical and sub-clinical) to ICD-9 Diagnoses supported by diagnostic, radiographic and/or MRI findings where clinically indicated.
  Other Names: Musculoskeletal Disorder Reporting Tool

SUMMARY:
To administer the MSDR® (Musculoskeletal Disorder Reporting) instrument to document the musculoskeletal profile of patients with chronic low back pain, a prospective, non-randomized, multicenter treatment trial

ELIGIBILITY:
Inclusion Criteria:

* Must have Informed Consent Signed
* Lumbar Disc Herniations under 5mm without Sequestered Fragments
* Lumbar Disc Bulging
* Lumbar Degenerative Disc Disease (mild and moderate severity)
* Non-pregnant Females and Males suffering from Chronic Low Back Pain from 18 to 65 years of age
* Segmental Dysfunction Secondary to Dyskinesia
* Unresolved Nerve Entrapment Syndrome
* Patients must be able to comply with study protocol
* Joint Fixation Syndrome
* Premenopausal Female Patients, excluding patients who have undergone a hysterectomy, oophorectomy, or tubal ligation, must have one of the following methods of contraception and must have a negative serum or urine b-HCG pregnancy test performed within 48 hours before initiating protocol specified treatment.

Exclusion Criteria:

* Contraindications to Spinal Manipulative Therapy
* Lumbar Canal Stenosis resulting in significant neurological comprimise
* Any Spinal Cord Compression resulting in significant neurological comprimise
* Cauda Equina Syndrome
* Infection
* Osteomyelitis

  ->65 years of age
* History of Back or Neck Surgery
* Acute Arthritis
* Signs or Symptoms of Arterial Aneurysm
* History of Active Cancer with Bone Metastasis
* Widespread Staphyloccal and/or Strepococcal Infection
* Acute Gout
* Serious unstable medical illness such as cardiovascular, renal, respiratory, endocrine, gastrointestinal, or psychiatric.
* Unstable Spondylosis, Spondylolisthesis, or Spondylolysis
* Prior adverse experience with Spinal Manipulation Therapy
* Uncontrolled Diabetic Neuropathy
* Gonorreal Spinal Arthritis
* Tuberculosis to the Bone
* Maligancy with Metatasis to Bone
* Excessive Spinal Osteoporosis
* Osteomalacia
* Ankylosis
* Syphlitic Articular or Peri-Articular Lesions
* Active Low Back Injury Resulting from a Motor Vehicle Accident or Work Related Injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-08 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
To document the musculoskeletal profile of patients with low back pain | 1 year

SECONDARY OUTCOMES:
To determine if a particular lower back diagnosis or MSDR® score can predict which patients will respond particularly well to the DRX9000™ treatment protocol and spinal manipulative therapy. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eric K Groteke, DC, Study Chair — MedAppraise, Inc.; Luis Crespo, MD, Principal Investigator — Crespo and Associates; Mark Scinico, MD, Study Director — Concentra; Damon J Stafford, DC, Principal Investigator — Back2Life of Florida, Inc.
Locations (1):
- Back2Life of Florida, Inc., Clearwater, Florida, United States

REFERENCES:
- See also: MSDR — http://www.medappraise.com